CLINICAL TRIAL: NCT04338906
Title: Evaluation of the Efficacy and Safety of Camostat Mesilate + Hydroxychloroquine Combination Therapy in Hospitalized Patients With Moderate COVID-19 Infection
Brief Title: Combination Therapy With Camostat Mesilate + Hydroxychloroquine for COVID-19
Acronym: CLOCC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of public funding; planned control arm with Hydroxychloroquine treatment showed out as not being standard of care anymore as time evolved.
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Goethe University (Other); St. Georg Hospital Leipzig, Germany (Unknown); Hospital Schwabing Munich, Germany (Unknown); Missioklinik, Wuerzburg, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOCC-2020
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: COVID
Keywords: Camostat; Hydroxychloroquine; Moderate COVID-10
MeSH Terms: interventions — camostat; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Evaluation of the efficacy and safety of hydroxychloroquine + camostat combination therapy in comparison to hydroxychloroquine + placebo in hospitalized patients with moderate COVID-19 infection, CLOCC-Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camostat + Hydroxychloroquine (Experimental): Subjects will receive Camostat (400 mg tid) + hydroxychloroquine (400 mg bid day1, 200 mg bid d2-d7)
  Interventions: Drug: Camostat Mesilate; Drug: Hydroxychloroquine
- Placebo + Hydroxychloroquine (Active Comparator): Subjects will receive placebo (tid) + hydroxychloroquine (400 mg bid day1, 200 mg bid d2-d7)
  Interventions: Drug: Placebo; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Camostat Mesilate — 400 mg tid, d1-d7
  Arms: Camostat + Hydroxychloroquine
Drug: Placebo — Instead of Camostat Mesilate, tid, d1-d7
  Arms: Placebo + Hydroxychloroquine
Drug: Hydroxychloroquine — 400 mg bid on day 1, 200 mg bid d2-d7

SUMMARY:
Evaluation of the efficacy and safety of hydroxychloroquine - camostat combination therapy in hospitalized patients with moderate COVID-19 infection, CLOCC-Trial Primary Objectives: The primary objective of this study is to demonstrate, that a combination therapy of hydroxychloroquine and camostat (Foipan®) is superior to hydroxychloroquine + placebo in participants with moderate COVID-19.

DETAILED DESCRIPTION:
The ongoing pandemic with the novel coronavirus (SARS-CoV-2) poses a massive threat to public health. SARS-CoV-2 is highly contagious and may lead to severe acute respiratory distress syndrome in affected individuals. No therapeutic intervention has yet been approved for COVID-19, and initial interventional studies with single agents showed only minimal improvement in outcome or were not convincing in design. Therefore, the CLOCC trial will evaluate the efficacy and safety of a combination therapy consisting of hydroxychloroquine, which was used already as single agent with some effect, together with camostat mesylate in hospitalized patients with moderate COVID-19 infection. The rationale for this combination therapy stems from the observation that hydroxychloroquine interferes with viral entry and replication through several mechanisms including changes in endosomal pH and in glycosylation of the ACE2 receptor, which serves as entry receptor for SARS-CoV-2. Camostat acts as inhibitor of the host cell serine protease TMPRSS2, which is needed to prime the viral S protein for cell entry. Participants will be recruited in a total of 6 German centers, and the trial will be randomized (1:1) and enrolled in either the hydroxychloroquine + placebo or the hydroxychloroquine + camostat arm (7-day treatment). The trial will be carried out in a double-blinded fashion. The primary efficacy outcome is the number of patients discharged by day 14 (status 1 and 2 of a 7-point ordinal clinical status scale). Several secondary outcomes regarding efficacy but also safety will be evaluated. Exploratory endpoints include analysis of viral titers and the emergence of viral resistance in response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age with SARS-CoV-2 infection confirmed by PCR before randomization
* Willing and able to provide written informed consent
* Hospitalized and requiring medical care for COVID-19, (status 3 or 4 of 7-point ordinal clinical status scale)
* SpO2 ≥93% on room air
* Evidence of pulmonary infiltrate on chest X ray/and or CT scan

Exclusion Criteria:

* Age <18 years old
* Pregnant or breast feeding
* Inability to take oral medication
* Inability to provide informed written consent
* Known hypersensitivity towards 4-aminoquinolines, e.g. hydroxychloroquine and/or camostat
* Use of hydroxychloroquine, chloroquine and or camostat within 6 months prior to baseline
* Patients with known retinopathy or macular degeneration Patients with known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Prolonged QTc-interval in baseline ECG (>500 ms)
* Concomitant medication associated with QTc-interval prolongation, which cannot be withdrawn prior to study drug administration
* Major comorbidities, possibly leading to increased unwanted side effects of study drugs:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Not hospitalized | day 14 from baseline

SECONDARY OUTCOMES:
Time to improvement of 2 categories from admission on a 7-point ordinal scale | day 14
Proportion of participants in each group with normalization of fever | day 7 and day 14
Proportion of participants in each group with oxygen saturation > 94% on room air for >24h | day 7 and day 14
Time to fever normalization (if febrile at baseline) | within 14 days
Time to first negative SARS-CoV-2 PCR in NP swap (if pos. at baseline) | within 14 days
Time to first negative SARS-CoV-2 PCR in lower respiratory tract specimens (sputum, bronchoalveolar lavage, tracheal aspirate) (if positive at baseline) | within 14 days
Duration of oxygen therapy | within 28 days
Proportion of participants in each group with need for mechanical ventilation | within 28 days
Duration of hospitalization | within 28 days
All cause mortality | day 28

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 Months after publication
Access Criteria: Open